CLINICAL TRIAL: NCT07259083
Title: Long-term Correlation of Functional and Psychological Parameters for the Return-to-sport Decision After Anterior Cruciate Ligament Reconstruction
Brief Title: Psychological and Physiological Parameters for Return-to-sport After ACL Reconstruction
Acronym: ACL-RTS
Status: Recruiting | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: University of Salzburg (Other)
Responsible Party: Principal Investigator, Christian Mittermaier, M.D., Johannes Kepler University of Linz
Other Study IDs: Kepler Universitätsklinikum /
Record Dates: First submitted 2025-04-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: ACL Reconstruction
Keywords: ACL rupture; ACL reconstruction; Return to sport; ACL tear; Dynamometry
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants after ACL reconstruction: 1 to 4 years after ACL reconstruction, age: 18 - 50 years, physically active

SUMMARY:
Injuries to the anterior cruciate ligament are common and are usually treated with reconstruction and subsequent rehabilitation. Many people succeed in return to sport (RTS), but not to the original level. Muscle strength factors can be assessed using isokinetic strength measurements, while the psychological readiness to return to sport can be assessed using the Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) questionnaire. In this study, isokinetic strength testing and psychological testing with the ACL-RSI questionnaire 1 to 4 years after ACL reconstruction will be assessed. The study will be conducted at the Institute of Physical Medicine & Rehabilitation at the Kepler University Hospital. The Biodex System Pro™, a medical device for measuring and training muscle strength, will be used for the isokinetic measurements. The research question is as follows: Is there a correlation between the results of the ACL RSI questionnaire and the results of isokinetic strength testing on the Biodex System 4 Pro™ in test subjects following ACL reconstruction?

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral ACL reconstruction 1 to 4 years prior testing
* Physically active
* 18-50 years
* Medical approval for maximum loads

Exclusion Criteria:

* Bilateral Knee injury
* Pregnancy
* Acute pain (VAS ≥ 3)
* Extremely limited mobility
* Extreme joint instability
* Acute injuries
* Inflammation
* Fever

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Physically active adults who underwent unilateral ACL reconstruction 1 to 4 years ago
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Peak torque (Nm) - Isokinetic dynamometry (Biodex System 4) | Day 1 (1 to 4 years after ACL reconstruction)
  The isokinetic dynamometer measures concentric strength in extension and flexion.
  Isokinetic strength testing at a ROM (range of motion) of 0-90° knee flexion at 3 different speeds. Test protocol at angular velocities of 60°/sec, 180°/sec and 240°/sec.
ACL-RSI questionnaire (Anterior Cruciate Ligament-Return to Sport after Injury) | Day 1 (1 to 4 years after ACL reconstruction)
  The ACL-RSI is a measure of psychological readiness to return to sport. It contains 12 questions and examines 3 components related to readiness to return to sport: emotions (5 questions), confidence in one's own performance (5 questions) and risk assessment (2 questions). The questions relate to the psychological effects of returning to sport. The respondents answer each question by giving their assessment in steps of ten on a Likert scale from 0 to 100 points. Low scores indicate a negative psychological assessment and high scores indicate a positive psychological assessment. The cut-off value for distinguishing between returnees and non-returnees is 51.3 points. A German version of the questionnaire is used.

SECONDARY OUTCOMES:
Isokinetic dynamometry (Biodex System 4) | Day 1 (1 to 4 years after ACL reconstruction)
  The isokinetic dynamometer measures concentric strength in extension and flexion including following parameters:
  Average peak torque (Nm), time to peak torque (sec), angle of peak torque (deg), torque at 30°, torque at 0.18 seconds, max. repetitions to total work, work/body weight, total work, work first third, work last third, work fatique, avg. power, acceleration time (msec), ROM (range of motion, deg), agonist/antagonist ratio (%), hamstring/quadriceps (H/Q) ratio, LSI (limb symmetry index)
  Isokinetic strength testing at a ROM of 0-90° knee flexion at 3 different speeds. Test protocol at angular velocities of 60°/sec, 180°/sec and 240°/sec.
Sports activity | Day 1
  Sports activity before and after surgery in minutes/week

OTHER OUTCOMES:
Time since ACL surgery | Day 1
  Time in months since ACL surgery
Height | Day 1
  Height of the participant in cm
Weight | Day 1
  Weight of the participant in kg
Body Mass Index | Day 1 (1 to 4 years after ACL reconstruction)
  Relation of body weight to the square of body height
Age | Day 1
  Age of the participant in years

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Clinic, Dept. of Physical Medicine & Rehabilitation, Linz, Austria

IPD SHARING:
Plan to Share IPD: No